CLINICAL TRIAL: NCT07170371
Title: Patient Education Program for Individuals With Rheumatoid Arthritis: A Randomized Controlled Trial
Brief Title: Patient Education and Rheumatoid Arthritis
Acronym: PE and RA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hassan II University (Other)
Responsible Party: Principal Investigator, Abdelaaziz Bounabe, Dr BOUNABE ABDELAAZI, Hassan II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D/2025/HASSANII/54
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-09

CONDITIONS: Rheumatoid Arthritis
Keywords: patient education
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two parallel groups. One group will receive a culturally adapted patient education program in addition to usual medical care, while the other group will receive usual care alone. The two groups will be followed for 6 months, with comparative evaluation of outcomes related to self-management and quality of life.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient education Group (Experimental): A culturally adapted patient education program designed for individuals with rheumatoid arthritis. The program was developed through a structured needs assessment and based on established health behavior theories. It includes five core modules delivered over six months: understanding rheumatoid arthritis, monitoring disease activity, treatment strategies, nutrition, and stress management. Sessions combine group workshops and individual support, with interactive materials and practical exercises. The program aims to strengthen patients' knowledge, self-management skills, and quality of life compared to usual care.
  Interventions: Other: patient education
- Usual care Group (Active Comparator): patients will receive usual care only
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: patient education — A culturally adapted patient education program designed for individuals with rheumatoid arthritis. The program was developed through a structured needs assessment and based on established health behavior theories. It includes five core modules delivered over six months: understanding rheumatoid arthritis, monitoring disease activity, treatment strategies, nutrition, and stress management. Sessions combine group workshops and individual support, with interactive materials and practical exercises. The program aims to strengthen patients' knowledge, self-management skills, and quality of life compared to usual care.
  Arms: Patient education Group
Other: Usual Care — patients will receive usual care only
  Arms: Usual care Group

SUMMARY:
The goal of this clinical trial is to learn if a culturally adapted patient education program can help people with rheumatoid arthritis (RA) manage their disease and improve their quality of life. The main questions it aims to answer are:

* Does the program improve patients' knowledge, self-management skills, and confidence in dealing with RA?
* Does it lead to better quality of life and treatment adherence compared to usual care?

Participants will:

* Join group sessions and individual activities focused on RA education, self-care, and stress management
* Take part in the program for 6 months, with regular follow-up visits
* Complete questionnaires about symptoms, daily activities, and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) diagnosed with rheumatoid arthritis according to ACR/EULAR 2010 classification criteria
* Stable pharmacological treatment for at least 3 months prior to enrollment
* Ability to participate in group sessions and complete questionnaires
* Provided written informed consent

Exclusion Criteria:

* Diagnosis of other systemic autoimmune or inflammatory rheumatic diseases (e.g., lupus, psoriatic arthritis)
* Severe comorbidities that may interfere with participation (e.g., advanced heart failure, uncontrolled psychiatric illness)
* Cognitive impairment or language barrier preventing comprehension of the program
* Participation in another structured patient education program within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
AIMS2 Quality of life | Baseline to 6 months after randomization
  Change in health-related quality of life among participants, measured using validated patient-reported questionnaires (AIMS2) to assess physical, emotional, and social domains. The focus is on improvement in self-reported well-being and daily functioning.

SECONDARY OUTCOMES:
DAS-28 | Baseline to 6 months after randomization
  Change in disease activity, assessed by the Disease Activity Score 28 (DAS28), including tender/swollen joint counts, ESR/CRP levels, and patient global assessment
ASES | Baseline to 6 months after randomization
  Change in patient self-efficacy for managing rheumatoid arthritis, assessed with the Arthritis Self-Efficacy Scale (ASES), covering pain, function, and other disease-related aspects.
MARS | Baseline to 6 months after randomization
  Change in treatment adherence measured by the Medication Adherence Rating Scale (MARS), focusing on consistency of drug intake and attitudes toward treatment.
BDI | Baseline to 6 months after randomization
  Change in depressive symptoms measured by the Beck Depression Inventory (BDI), and in perceived stress using standardized self-report tools

CONTACTS AND LOCATIONS:
Locations (1):
- university hospital IBN ROCHD, Casablanca, Morocco

IPD SHARING:
Plan to Share IPD: No